CLINICAL TRIAL: NCT03943628
Title: Families Preventing and Reducing Obesity Health Disparities in Hispanic Youth
Brief Title: Reducing Obesity Health Disparities in Hispanic Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Guillermo Prado, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20130195; R01MD007724 (NIH)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Overweight; Family Relations; Adolescent Behavior; Drug Use; Sexual Behavior
Keywords: prevention; Hispanic adolescents; obesity and overweightness; family functioning; sexual risk behavior
MeSH Terms: conditions — Overweight; Adolescent Behavior; Sexual Behavior; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Familias Unidas (Experimental): Consists of eight parent group sessions and four family sessions with the adolescent.
  Interventions: Behavioral: Familias Unidas
- Community Practice (Other): Consists of community practice.
  Interventions: Behavioral: Familias Unidas

INTERVENTIONS:
Behavioral: Familias Unidas

SUMMARY:
The proposed study will evaluate the efficacy of a family-based obesity prevention intervention in increasing physical activity and improving the quality of dietary intake among Hispanic Youth. Additional primary outcomes that will be examined include drug use and sexual risk behaviors. Secondary outcomes include examining the effects of family functioning and BMI. The knowledge expected to be gained in this study will have strong implications for prevention as well as contribute to the reduction of obesity-related health disparities seen in Hispanic youth.

DETAILED DESCRIPTION:
This study's aims are: AIM 1: To examine the relative efficacy of Familias Unidas, extended to target obesity, in increasing physical activity and improving the quality of dietary intake among overweight Hispanic youth and AIM 2: To examine whether and to what extent family functioning partially mediates the effects of Familias Unidas on physical activity and quality of dietary intake.

H1: Familias Unidas will be efficacious, compared to Community Practice, in increasing Hispanic youth's past moderate to vigorous physical activity over time.

H2: Familias Unidas will be efficacious, compared to Community Practice, in improving Hispanic youth's past quality dietary intake (defined as decreases in dietary intakes of sugar-sweetened beverages, fast foods, and increases in dietary intakes of fresh fruits and vegetables) over time.

H3: Familias Unidas' effects on youth's past day moderate to vigorous physical activity and youth's past quality dietary intake will be partially mediated by changes in family functioning over time.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Female and male adolescents of Hispanic immigrant origin, defined by at least one parent (or legal guardian/primary caregiver) born in a Spanish speaking country of the Americas.
2. Adolescent attending 7th or 8th grade at the time of the initial assessment (T1).
3. Adolescent living with an adult primary caregiver who is willing to participate in the study.
4. At T1, families must live within the catchment areas of the middle schools included in this study: Citrus Grove, Shenandoah Middle, Kinloch Park, Ponce de Leon, Rivera, South Miami, Glades, and Carver Middle Schools. All eight schools are located within a single school district, and have a population that is predominantly Hispanic (70% or greater across all three schools). Our staff has conducted studies with these schools for over 15 years (see letter of support from the Miami-Dade County Public School District), which collectively serve over 2,000 Hispanic 8th graders per year. We will be recruiting over three academic school years. Thus, we do not anticipate any barriers to recruiting the target sample size from the 6,000 Hispanic 8th graders (of which approximately 1800 are expected to be overweight) enrolled in these schools over the three academic years.
5. Adolescents must meet criterion for overweight (i.e. body mass index [BMI] > 85% adjusted for age and sex). We decided to select overweight youth for a number of reasons: (1) In our prior research with Familias Unidas, we have found that our intervention is most successful for more at- risk samples and less efficacious for universal samples (IOM, 2009) and (2) The needs of normal- weight (or underweight) youth may not be adequately or appropriately addressed by a family-based intervention targeting behavioral risk factors for obesity. For example, Whitlock and colleagues found that including normal-weight youth in research studies may induce individual and parental preoccupation with weight, weight management, and dietary and physical activity behaviors and, thus, have iatrogenic effects (Whitlock et al., 2005).

EXCLUSION CRITERIA:

(a) Family planning to move out of the catchment areas of the target schools during the 3 month intervention period, or out of the South Florida area during the two year follow-up phase of the study. (b) Parent or youth refuses to participate in the study.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Physical Activity Questionnaire | Baseline and 6-, 12-, 24- months post-baseline
  Change in moderate to vigorous physical activity over time
NHANES Dietary Screener Questionnaire (DSQ) | Baseline and 6-, 12-, 24- months post-baseline
  Change in quality dietary intake (decreases in dietary intakes of sugar-sweetened beverages, fast foods, and increases in dietary intakes of fresh fruits and vegetables) over time.

SECONDARY OUTCOMES:
BMI | Baseline and 6-, 12-, 24- months post-baseline
  Collection of raw BMI data for children and adults
Parenting Practices Questionnaire | Baseline and 6-, 12-, 24- months post-baseline
  Measure to assess parental investment
Parent-Adolescent Communication Scale | Baseline and 6-, 12-, 24- months post-baseline
  Measure to assess quality and content of communication. Items are measured on a scale from 1= Strongly disagree, 2=Moderately disagree, 3=Neither agree nor disagree, 4=Moderately agree and 5=Strongly agree. Higher values represent a better outcome. Sum scores are used to determine a total score
Drug Use (items from Monitoring the Future Survey) | Baseline and 6-, 12-, 24- months post-baseline
  Measure to assess frequency of adolescent drug use
Adolescent Sexual Risk Behaviors | Baseline and 6-, 12-, 24- months post-baseline
  Measure to assess adolescent sexual activity

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Prado, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perrino T, Brincks AM, Estrada Y, Messiah SE, Prado G. Reducing Screen-Based Sedentary Behavior Among Overweight and Obese Hispanic Adolescents Through a Family-Based Intervention. J Phys Act Health. 2022 Jul 7;19(7):509-517. doi: 10.1123/jpah.2022-0050. Print 2022 Jul 1. PMID 35894971
- [Derived] Kobayashi MA, Lee TK, St George SM, Lebron C, Dorcius D, Prado G, Messiah SE. Intergenerational cardiovascular disease risks among Hispanics living in the United States. Pediatr Obes. 2022 Apr;17(4):e12870. doi: 10.1111/ijpo.12870. Epub 2021 Nov 8. PMID 34751514
- [Derived] Fernandez A, Lozano A, Lee TK, Estrada Y, Messiah SE, Prado G. A Family-Based Healthy Lifestyle Intervention: Crossover Effects on Substance Use and Sexual Risk Behaviors. Prev Sci. 2021 Jul;22(5):602-608. doi: 10.1007/s11121-021-01220-z. Epub 2021 Mar 10. PMID 33689118
- [Derived] Prado G, Fernandez A, St George SM, Lee TK, Lebron C, Tapia MI, Velazquez MR, Messiah SE. Results of a Family-Based Intervention Promoting Healthy Weight Strategies in Overweight Hispanic Adolescents and Parents: An RCT. Am J Prev Med. 2020 Nov;59(5):658-668. doi: 10.1016/j.amepre.2020.06.010. Epub 2020 Oct 1. PMID 33011010